CLINICAL TRIAL: NCT02841384
Title: McConnell Patellar Taping in Static and Dynamic Postural Control of Women With Patellofemoral Pain Syndrome: Randomized Clinical Trial and Blind
Brief Title: McConnell Patellar Taping in Static and Dynamic Postural Control of Women With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, First investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mcconnelltaping
Record Dates: First submitted 2016-07-01; First posted 2016-07-22 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; postural balance; knee; physiotherapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group taping McConnell (Other): Taping patellar McConnell: Lateralization correction of the patella with self-adhesive rigid bandage Johnson® positioned lateral border of the patella to the medial condyle of the femur, allowing the lifting of the medial border of the patella and stretching of the knee lateral structures.
  Interventions: Other: taping patellar McConnell
- Group placebo taping (Other): Placebo taping through vertical application of patellar rigid taping, with the knee in flexion without medialization of the patella.
  Interventions: Other: Placebo taping

INTERVENTIONS:
Other: taping patellar McConnell — Taping patellar McConnell: Lateralization correction of the patella with self-adhesive rigid bandage Johnson® positioned lateral border of the patella to the medial condyle of the femur, allowing the lifting of the medial border of the patella and stretching of the knee lateral structures.
  Arms: Group taping McConnell
Other: Placebo taping — Placebo taping through vertical application of patellar rigid taping, with the knee in flexion without medialization of the patella.
  Arms: Group placebo taping

SUMMARY:
Introduction: Patellofemoral pain syndrome (PFPS) is related to the previous sore knee, change functionality and postural control deficits. One of the possibilities for pain control and better positioning of the patella is the rigid bandage patellar widely used by clinicians and researchers.

Objective: To evaluate the effect of rigid patellar bandage on postural control, pain and function in sedentary women with PFPS.

Methods: The sample will be composed of 30 volunteers, sedentary, between 18 and 55 years; randomized group Bandage Functional Rigid (n = 15) and Banding Placebo (n = 15). All fill the Personal Data Sheet, Visual analog scale Pain Questionnaire Previous Knee Pain Scale; and will be submitted to analysis of postural control (static and dynamic) and carry out the test and sit up in pre conditions and post application of the bandage.

Hypothesis: Expected to observe the effect of rigid patellar bandage in pain, function and postural control in sedentary women with PFPS.

DETAILED DESCRIPTION:
This is a randomized controlled trial and blind in the exercise area, postural control and biomechanics.

The subjects with a clinical diagnosis of PFPS will be allocated in two groups: PFPS group with rigid bandage patella (n = 15) and PFPS group with placebo (n = 15).

Procedures: The subjects with a clinical diagnosis of PFPS, will be forwarded to the evaluation protocols. The data collections will be held at University Hospital Physiotherapy Division of the State University of Londrina. Individuals respond to a questionnaire to characterize the sample, EVA and fill the patellofemoral disorders Scale (AKPS).

Data Collection Protocol: will be held to familiarize themselves with the equipment and tests to be used on the force platform and test sitting and standing, voluntary is inserted in one of the groups (PPS + B or PPS + P) through randomisation previously established by www.random.org and stored in opaque and sealed envelopes.

Following the participants carry out, random and drawn at the time way, the static and dynamic tests on the force platform:

Static: The volunteers will stay 30 seconds in one-leg position of the lower limb with pain with the knee flexed and contralateral suspended to about 90; the test will be performed three times, with one minute of sitting home. Participants will be instructed to keep aligned and torso upright during the test and stay as long as possible with most of the plantar region touching the ground. Will be targeted to fix the look upon in a pre-established and pasted on the wall point.

Dynamic Squat: The volunteers will perform three consecutive repetitions of squat exercise, controlled between about 0 ° to 45 ° of knee flexion in the lower limb with pain. The contralateral leg should be suspended and flexed to 90 °, the activity will be performed three times, with one minute rest in the sitting position between each repetition. Participants will be instructed to keep aligned and torso upright during the test and stay as long as possible with most of the plantar region touching the ground. Will be targeted to fix the look upon in a pre-established and pasted on the wall point.

Dynamic Up and Down Stairs: The force platform will be positioned at 20 cm from the ground on a wooden structure. The front is combined with a second step, also with 20 cm high from the first step, simulating a staircase with two steps of 20 cm each. Voluntary perform the functional activity of climbing the two steps, starting the first step with the leg with pain to support the platform. The activity will be carried out three consecutive times, with rest of a seated minute, and then the voluntary hold the decline in two steps, with lower limb support with pain on the platform, also performed by three consecutive times.

The average of the three repetitions of each activity (static and dynamic) will be used for postural control analysis (COP parameters) for each variable to be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of patellofemoral dysfunction issued by a specialist orthopedic knee and provide anterior knee pain of 3 or more on the Visual Analogue Scale (VAS) for a minimum of 8 weeks prior to evaluation;
* Previous retropatellar pain or knee, for at least 3 of the following: up / down stairs, squatting, running, kneeling, sitting for long periods and insidious onset of symptoms unrelated to trauma.

Exclusion Criteria:

* History of severe / traumatic knee injury, surgery history in the locomotor system;
* Patellar luxation history; clinical evidence of meniscus injury; ligamentous instability; patellar tendinitis.
* Presence of neurological, cardiovascular or rheumatologic diseases; pregnancy; diabetes,
* Abnormal sensitivity in the plantar;
* Medication and / or therapy in the last six months and hypersensitivity or allergy to tape.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01; Primary Completion 2016-12-30 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
change the balance after the intervention by force platform | before and immediately after the intervention
  It will be measured the oscillations through various force platform variables before and after the intervention (taping or placebo, depending on the group) to see if there is change in the balance after the implementation of these interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, doctor, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- university hospital of the State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee SE, Cho SH. The effect of McConnell taping on vastus medialis and lateralis activity during squatting in adults with patellofemoral pain syndrome. J Exerc Rehabil. 2013 Apr;9(2):326-30. doi: 10.12965/jer.130018. Epub 2013 Apr 25. PMID 24278879
- [Result] Felicio LR, Masullo Cde L, Saad MC, Bevilaqua-Grossi D. The effect of a patellar bandage on the postural control of individuals with patellofemoral pain syndrome. J Phys Ther Sci. 2014 Mar;26(3):461-4. doi: 10.1589/jpts.26.461. Epub 2014 Mar 25. PMID 24707108